CLINICAL TRIAL: NCT04089319
Title: Acupuncture Combined With Mindfulness in the Context of Chronic Pain
Brief Title: Acupuncture Combined With Mindfulness: ACUMIND
Acronym: ACUMIND
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 prevented us from recruiting additional participants.
Sponsor: University of Utah (Other)
Collaborators: Huntsman Cancer Institute (Other)
Responsible Party: Principal Investigator, Lisa J Taylor-Swanson, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 00108827
Record Dates: First submitted 2019-09-10; First posted 2019-09-13 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Acupuncture; Mindfulness; Interoceptive Awareness
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture + mindfulness (Experimental): Participants will receive acupuncture treatment for chronic pain. After acupuncture needles have been inserted, participants will listen to a 15-minute mindfulness recording followed by music for 30 minutes. Acupuncture needles will then be removed.
  Interventions: Other: Mindfulness recording
- Acupuncture control (Other): Participants will receive acupuncture treatment for chronic pain. After acupuncture needles have been inserted, participants will listen music for 45 minutes. Acupuncture needles will then be removed.
  Interventions: Other: Music recording

INTERVENTIONS:
Other: Music recording — Participants will listen to music for 45 minutes while they rest with acupuncture needles in place.
  Arms: Acupuncture control
Other: Mindfulness recording — Participants will listen to a recording of mindfulness for 15 minutes and then listen to music for 30 minutes while they rest with acupuncture needles in place.
  Arms: Acupuncture + mindfulness

SUMMARY:
This study aims to gather preliminary data regarding acupuncture and mindfulness in the treatment of chronic pain.

DETAILED DESCRIPTION:
Neither acupuncture nor mindfulness have been studied with respect to chronic pain in an outpatient integrative health (IH) oncology clinic in the USA. Likewise, the combination of acupuncture and mindfulness combined as not been studied. Given that both acupuncture and mindfulness have demonstrated some analgesic relief in an acute pain setting, each merit study for pain relief in an outpatient setting.

The investigators are evaluating the impact of two different acupuncture approaches for patients reporting chronic pain. Acupuncture will be provided by a Licensed Acupuncturist for patients reporting chronic pain. Participants will be randomized to one of two treatments - acupuncture as usual or acupuncture plus mindfulness.

The investigators will collect data regarding chronic pain, interoceptive awareness, emotion regulation, and acceptability. The study is open to participants with any etiology and any location of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient is age 18 or older.
* Patient is experiencing pain (rated ≥3 on a 0-10 scale) lasting for three or more months.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* ONLY FOR THOSE WITH A DIAGNOSIS OF CANCER: ECOG status of 0 (asymptomatic), 1 (symptomatic but completely ambulatory) or 2 (symptomatic, <50% in bed during the day).

Exclusion Criteria:

* Patient has received 5 or more acupuncture treatments in the last 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Questions Regarding Pain and Other Symptoms | 2 months
  A questionnaire regarding pain as well as physical and mental awareness. A Likert scale 0-10 is used, where 0 is classified as "not at all" and 10 is classified "very much." Higher values are a worse outcome with questions 7-9 reverse scored.

SECONDARY OUTCOMES:
Nondual Awareness Dimensional Assessment | 2 months
  A questionnaire regarding nondual awareness. Scored on a 10-point Likert scale (1=Not at all, 10=Very Much), higher values are a better outcome.
State Difficulties in Emotion Regulation Scale | 2 months
  A questionnaire regarding emotional awareness. Scored on a 5 point Likert scale (1=not at all, 5=completely), higher values are a better outcome.
Sensation Manikin | 2 months
  A map of the body used to identify and measure areas of pleasant and unpleasant sensations.
Retrospective Chart Review | 3 month
  To discover pain medications taken by participant in the last 90 days, including opioid dose (to be converted into morphine milligram equivalent, MME).
State Multidimensional Assessment of Interoceptive Awareness-2 | 2 months
  A questionnaire regarding interoceptive awareness. Scored on a 6-point Likert scale (0=never, 5=always), higher values are a better outcome.
Acupuncture Questions | 2 months
  A questionnaire regarding changes in sensations experienced during the AT. This is scored on a 6-point Likert scale (0=not at all, 5=to all the time/every location), higher values are a better outcome.
Acceptability Questions | 1 day
  A questionnaire regarding the acceptability of the AT. This is scored on a 5 point Likert scale (1=completely disagree, 5=completely agree), higher values are a better outcome.
Qualitative Inquiry | 1 day
  A questionnaire regarding experiences during the AT. This consists of free response questions.
Qualitative Interoceptive Awareness and Emotional Regulation | 1 day
  A questionnaire regarding changes experienced since AT. This consists of open ended text questions.
Quantitative questions | 1 day
  A questionnaire regarding overall health since AT. Questions 1-3 are scored on a Likert scale 0-10 is used where 0 is classified as "not at all" and 10 is classified "very much" with higher values indicating a better score and question 1 is reverse scored. Questions 4-8 are measured on a 5 point Likert scale (1=not at all, 5=completely) with higher values indicating a better outcome. Question 9 is scored on a 1-5 Likert scale with lower values indicating a better outcome. Questions 10-19 are scored on a 3 point Likert scale with higher values indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Taylor-Swanson, PhD, MAcOM, Principal Investigator — University of Utah College of Nursing; Annie Budhathoki, LAc, DAOM, Study Director — Huntsman Cancer Institute; Eric Garland, Study Director — University of Utah College of Social Work, Huntsman Cancer Institute; Shelley White, PhD(C), MSW, Study Director — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Individual data is not useful data at this stage.

REFERENCES:
- [Background] Rainville P. Brain mechanisms of pain affect and pain modulation. Curr Opin Neurobiol. 2002 Apr;12(2):195-204. doi: 10.1016/s0959-4388(02)00313-6. PMID 12015237
- [Background] Lau MA, Bishop SR, Segal ZV, Buis T, Anderson ND, Carlson L, Shapiro S, Carmody J, Abbey S, Devins G. The Toronto Mindfulness Scale: development and validation. J Clin Psychol. 2006 Dec;62(12):1445-67. doi: 10.1002/jclp.20326. PMID 17019673
- [Background] Lang PJ, Davis M. Emotion, motivation, and the brain: reflex foundations in animal and human research. Prog Brain Res. 2006;156:3-29. doi: 10.1016/S0079-6123(06)56001-7. PMID 17015072
- [Background] Froeliger B, Mathew AR, McConnell PA, Eichberg C, Saladin ME, Carpenter MJ, Garland EL. Restructuring Reward Mechanisms in Nicotine Addiction: A Pilot fMRI Study of Mindfulness-Oriented Recovery Enhancement for Cigarette Smokers. Evid Based Complement Alternat Med. 2017;2017:7018014. doi: 10.1155/2017/7018014. Epub 2017 Mar 8. PMID 28373890
- [Background] Goldberg DS, McGee SJ. Pain as a global public health priority. BMC Public Health. 2011 Oct 6;11:770. doi: 10.1186/1471-2458-11-770. PMID 21978149
- [Background] Koleva D, Krulichova I, Bertolini G, Caimi V, Garattini L. Pain in primary care: an Italian survey. Eur J Public Health. 2005 Oct;15(5):475-9. doi: 10.1093/eurpub/cki033. Epub 2005 Sep 8. PMID 16150816
- [Background] Mantyselka P, Kumpusalo E, Ahonen R, Kumpusalo A, Kauhanen J, Viinamaki H, Halonen P, Takala J. Pain as a reason to visit the doctor: a study in Finnish primary health care. Pain. 2001 Jan;89(2-3):175-80. doi: 10.1016/s0304-3959(00)00361-4. PMID 11166473
- [Background] Breivik H, Cherny N, Collett B, de Conno F, Filbet M, Foubert AJ, Cohen R, Dow L. Cancer-related pain: a pan-European survey of prevalence, treatment, and patient attitudes. Ann Oncol. 2009 Aug;20(8):1420-33. doi: 10.1093/annonc/mdp001. Epub 2009 Feb 24. PMID 19244085
- [Background] Grissa MH, Baccouche H, Boubaker H, Beltaief K, Bzeouich N, Fredj N, Msolli MA, Boukef R, Bouida W, Nouira S. Acupuncture vs intravenous morphine in the management of acute pain in the ED. Am J Emerg Med. 2016 Nov;34(11):2112-2116. doi: 10.1016/j.ajem.2016.07.028. Epub 2016 Jul 20. PMID 27475042
- [Background] Vickers AJ, Cronin AM, Maschino AC, Lewith G, MacPherson H, Foster NE, Sherman KJ, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for chronic pain: individual patient data meta-analysis. Arch Intern Med. 2012 Oct 22;172(19):1444-53. doi: 10.1001/archinternmed.2012.3654. PMID 22965186
- [Background] Merskey H, Bogduk N. Classification of Chronic Pain: Descriptions of Chronic Pain Syndromes and Definitions of Pain Terms. 2nd ed. Seattle, WA, USA: International Association for the Study of Pain (IASP) Press; 1994.
- [Background] Lavender JM, Tull MT, DiLillo D, Messman-Moore T, Gratz KL. Development and Validation of a State-Based Measure of Emotion Dysregulation. Assessment. 2017 Mar;24(2):197-209. doi: 10.1177/1073191115601218. Epub 2016 Jul 27. PMID 26297011
- [Background] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087
- [Background] Hanley AW, Nakamura Y, Garland EL. The Nondual Awareness Dimensional Assessment (NADA): New tools to assess nondual traits and states of consciousness occurring within and beyond the context of meditation. Psychol Assess. 2018 Dec;30(12):1625-1639. doi: 10.1037/pas0000615. Epub 2018 Jul 30. PMID 30058824
- [Background] Hanley AW, Garland EL. Mapping the Affective Dimension of Embodiment With the Sensation Manikin: Validation Among Chronic Pain Patients and Modification by Mindfulness-Oriented Recovery Enhancement. Psychosom Med. 2019 Sep;81(7):612-621. doi: 10.1097/PSY.0000000000000725. PMID 31246748
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914